CLINICAL TRIAL: NCT03771092
Title: CONTROLLED RANDOMIZED PILOT STUDY TO COMPARE THE EFFICACY OF DIFFERENT IRON FORMULATIONS: SUCROSOMAL FERRIC PYROPHOSPHATE, SUNACTIVE Fe AND INTRAVENOUS FERRIC GLUCONATE
Brief Title: Comparing the Efficacy of Different Iron Formulations: Sucrosomal Ferric Pyrophosphate, SunActive®Fe and Intravenous Ferric Gluconate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Salvatore Corrao, MD, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREAM-IRON
Record Dates: First submitted 2018-11-06; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron; Iron Deficiency Anemia; Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patients with non-severe anemia treated with SunActive®Fe (Experimental): Patients with non-severe anemia Hb> 10 g/dl (Hb <12 g/dl for women and Hb <13 g/dl for men), treated with SunActive®Fe micronized
  Interventions: Dietary Supplement: SunActive®Fe
- Patients with non-severe anemia treated with Lipofer® (Experimental): Patients with non-severe anemia Hb> 10 g/dl (Hb <12 g/dl for women and Hb <13 g/dl for men), treated with Lipofer®
  Interventions: Dietary Supplement: Lipofer®
- Patients with severe anemia with Lipofer® (Experimental): Patients with severe anemia (Hb <10 g/dl) treated respectively with Lipofer®
  Interventions: Dietary Supplement: Lipofer®
- Patients with severe anemia with SunActive®Fe (Experimental): Patients with severe anemia (Hb <10 g/dl) treated respectively with SunActive®Fe micronized
  Interventions: Dietary Supplement: SunActive®Fe
- Patients with severe anemia with intravenous ferric gluconate (Experimental): Patients with severe anemia (Hb <10 g/dl) treated respectively with intravenous ferric gluconate according to departmental protocols
  Interventions: Dietary Supplement: Intravenous ferric gluconate

INTERVENTIONS:
Dietary Supplement: SunActive®Fe — SunActive® Fe is a colorless, odorless, tasteless iron fortifier in a powder form. This product is most commonly used to increase the amount of iron in food, beverage, and dietary supplement applications.
  Arms: Patients with non-severe anemia treated with SunActive®Fe; Patients with severe anemia with SunActive®Fe
Dietary Supplement: Lipofer® — Lipofer® is a micronized and microencapsulated source of iron, enhances the bioavailability of iron and does not taste metallic or oxidize unsaturated fats.
  Arms: Patients with non-severe anemia treated with Lipofer®; Patients with severe anemia with Lipofer®
Dietary Supplement: Intravenous ferric gluconate — Sodium ferric gluconate complex is an iron replacement product for treatment of iron deficiency anemia. The stable macromolecular complex is negatively charged at alkaline pH with an apparent molecular weight of 289,000 - 440,000 daltons on gel chromatography. It is composed of iron (III) oxide hydrate directly bonded to sucrose with a chelating gluconate function in a molar ratio of two iron molecules to one gluconate.
  Arms: Patients with severe anemia with intravenous ferric gluconate

SUMMARY:
The purpose of the study is to evaluate the effects of martial therapy, comparing different formulations, sucrosomal ferric pyrophosphate, SunActive®Fe micronized and ferric gluconate and different ways of administration, orally and intravenous, in subjects affected by sideropenic microcytic hypochromic anemia identified by the simultaneous presence of anemia, microcytosis and hypoferremia.

DETAILED DESCRIPTION:
Background: Iron deficiency anemia (IDA) still remains universally a worldwide problematics. Anemia is defined as a hemoglobin value <12.0 g/dL (7.45 mmol/L). Management of IDA is based on martial iron supplementation. The purpose of the study is to evaluate the effects of martial therapy, comparing different formulations, sucrosomal ferric pyrophosphate, SunActive®Fe micronized and ferric gluconate and different ways of administration, orally and intravenous, in subjects affected by sideropenic microcytic hypochromic anemia identified by the simultaneous presence of anemia, microcytosis and hypoferremia.

Trial Design, Methods and Findings: Clinical data from 106 outpatients (82.8% female and 17.2% male, mean age 50.4 years) were collected at Department of Internal Medicine, National Relevance and High Specialization Hospital Trust, ARNAS Civico-Di Cristina-Benfratelli, Palermo, Italy. The study envisaged five arms (2 + 3). At the first two arms were assigned patients with non-severe anemia Hb> 10 g/dl (Hb <12 g/dl for women and Hb <13 g/dl for men), treated with SunActive®Fe micronized or Lipofer®. At the other three arms were assigned patients with severe anemia (Hb <10 g/dl) treated respectively with SunActive®Fe micronized, Lipofer® or with intravenous ferric gluconate infusions according to departmental protocols. The followed methodology is defined in the PROBE project (acronym of Prospective Randomized Open Blinded End-point). The end points will be blinded with respect to the three treatments, as it will be the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of iron deficiency anemia, microcytic and hypochromic
* Age >18

Exclusion Criteria:

* Diagnosis of Celiac Disease
* Patients who refuse to sign the informed consent
* Clinically relevant cognitive Turbe
* Hemodynamic instability defined by the presence of low blood pressure SBP <100 FC> 100
* Dyspnea after modest effort worsening over the past 10 days
* Oxygen peripheral saturation values <94%
* Ischemic heart Recent and / or lower limbs
* Acute conditions with subacute or at recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
HB | Three months
  Mean change of hemoglobin concentration at three months

IPD SHARING:
Plan to Share IPD: No